CLINICAL TRIAL: NCT04876560
Title: The Use of Clinical Decision Support Systems (CDSS) to Provide Nutritional Care to Breast Cancer Patients During the COVID-19 Pandemic: a Randomised Controlled, Pilot Trial
Brief Title: Implementation of a CDSS in Oncology Patients During COVID-19
Acronym: CDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iaso Maternity Hospital, Athens, Greece (Other)
Collaborators: Harokopio University (Other)
Responsible Party: Principal Investigator, Panos Papandreou, PharmD, Iaso Maternity Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 31052019
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Obesity; Cardiovascular Disease Other
Keywords: decision support systems; breast cancer; Mediterranean diet; obesity; cardiovascular disease; quality of life
MeSH Terms: conditions — Breast Neoplasms; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSS (intervention) group (Active Comparator): Personalised nutritional advice: daily dietary programme with specific meals, products, recipes, food portions (in grams) based on the Meditteranean diet together with physical activity guidelines, all generated by a food database clinical decision support system (CDSS). Scheduled phone interviews every 15 days with the appointed dieticians assisted nutritional and lifestyle consultation.
  Interventions: Other: Application of CDSS to provide nutritional care in breast cancer patients from home
- Control group (Other): General lifestyle advice: based on the updated "American Cancer Society Guidelines on Nutrition and Physical Activity for Cancer Prevention" via scheduled phone interviews every 15 days.
  Interventions: Other: General lifestyle advice to breast cancer patients by phone

INTERVENTIONS:
Other: Application of CDSS to provide nutritional care in breast cancer patients from home — A personalised dietary plan was implemented by the CDSS. The CDSS estimated body mass index (BMI) and Total daily Energy Expenditure (TEE) according to individual's incorporated data. For overweight and obese patients, the CDSS produced a hypocaloric diet, in which daily energy intake was less than TEE by approximately -500 kcal/day. Nutrient distribution was in line with the Mediterranean dietary pattern. Patients received individual login passwords to CDSS allowing access to their personal profile from home. During the trial, patients were instructed to record food diaries in the CDSS every week, which were also made available to the dieticians. Visiting the CDSS, patients had the opportunity to track their progress e.g. monitoring goals of body weight, physical activity, consumption of fruits, vegetables, legumes.
  Arms: CDSS (intervention) group
Other: General lifestyle advice to breast cancer patients by phone — General lifestyle guidelines were provided by phone and food diaries were sent via emails.
  Arms: Control group

SUMMARY:
The present randomised controlled trial aimed to investigate the effectiveness of a clinical decision support system (CDSS) in assisting clinicians to apply nutritional care to breast cancer (BC) patients during the COVID-19 pandemic in Greece. Adult BC women (stages I-IIIA) who underwent mastectomy followed by hormone therapy were randomly assigned either to the Control group, receiving general nutritional advice, or the Intervention (or CDSS) group, in whom a personalised nutritional programme based on the Mediterranean diet together with physical activity guidelines were provided, all produced by CDSS. Medical and dietary history, anthropometrics, biochemical indices and quality of life characteristics were assessed both at baseline and at the end of the study (3 months).

DETAILED DESCRIPTION:
In this two-armed, single center, randomised controlled 3-month trial, simple randomisation was followed and the randomisation sequence was computer generated by an independent statistician. Blinding of the allocated treatment was maintained to the data analyst and was exposed only after the assessment of outcomes. Adult women (≥ 18 years of age) with histological evidence of primary invasive breast cancer (BC) at stages I-IIIA, who underwent mastectomy followed by antiestrogen therapy, were enrolled in the study. Additional criterion was the ability to ambulate independently, that corresponded to scoring 0 or 1 of the Eastern Cooperative Oncology Performance Status.

At baseline before the start of the trial, each enrolled participant completed a personal interview with the appointed dieticians. In the Intervention group (or CDSS group), patients received a personalised daily dietary plan (specific meals, products, recipes, food portions in grams) based on the Meditteranean diet together with physical activity guidelines, all generated by a newly developed clinical decision support system (CDSS). During the trial, BC women were instructed to record food diaries in the CDSS every week (2 weekdays and 1 weekend day), which were also made available to the dieticians. Visiting the CDSS, patients had the opportunity to track their progress e.g. monitoring goals of body weight, physical activity, consumption of fruits, vegetables, legumes. Regular phone interviews were scheduled on 15-day basis to assist nutritional and lifestyle consultation, while unexpected phone calls were made to receive 24-hour dietary records.

The Control arm received general lifestyle guidelines based on the updated "American Cancer Society Guidelines on Nutrition and Physical Activity for Cancer Prevention" via scheduled phone interviews every 15 days. Food diaries of each week (2 weekdays and 1 weekend day) were sent via emails and unexpected phone calls were made to receive 24-hour dietary records as well.

The appointed oncologist recorded medical history, including general information (age, sex, smoking) and disease specific data (i.e. cancer stage, type, age of diagnosis, symptoms and complications, and treatment). All assessments were carried out at the beginning and the end of the study (3 months). Body weight and body fat mass were measured with the method of Air Displacement Plethysmography. Dietary intake was evaluated using a semi-quantitative Food Frequency Questionnaire (FFQ), food diaries and 24h-recall records. The degree of Mediterranean diet adherence was estimated by the MedDiet score. The investigators also assessed performance status and physical activity, as well as quality of life and psychological distress by validated questionnaires. Our hypothesis was that the CDSS could be a useful means to provide nutritional care to BC patients ameliorating adherence to Mediterranean diet and the overall quality of life, during challenging periods like the COVID-19 pandemic.

ELIGIBILITY:
Inclusion criteria:

* Adult women (≥ 37 years of age);
* histological evidence of primary invasive breast cancer at stages I-IIIA;
* treatment: mastectomy followed by antiestrogen therapy;
* the ability to ambulate independently, that corresponded to scoring 0 or 1 of the Eastern Cooperative Oncology Performance Status

Exclusion criteria:

* Any other malignancy ≤ 5 years;
* co-existing medical conditions (e.g., obstructive ileus) that would interfere with the study protocol;
* malabsorption; serious chronic diseases (e.g. advanced heart, liver or renal failure, congenital metabolic diseases);
* active infection;
* severe psychiatric illness;
* alcoholism or drug use;
* vitamin or inorganic supplement use ≤ 6 months prior to screening;
* vegan or macrobiotic diet ≤ 5 years prior to screening;
* using weight loss medications.

Ages: 37 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
change in the Mediterranean diet adherence | 3 months
  detection of signrificantly greater adherence to Mediterranean diet in the CDSS (intervention) group compared to control group at study endpoint; assessed by the "MedDiet score"; scoring values 0 - 55; higher scores indicate greater adherence to the Mediterranean diet
change in "Global health, quality of life" score | 3 months
  detection of significantly higher "Global health, quality of life" score in the CDSS (intervention) group compared to control group at study endpoint; assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 items (EORTC QLQ-C30); scoring values 0 - 100; higher scores indicate greater overall quality of life

SECONDARY OUTCOMES:
alterations in the amount of daily intake of nutrients | 3 months
  detection of statistically significant differences in the amount of daily dietary intakes of fibers, monounsaturated fatty acids, saturated fatty acids, vitamin C between the CDSS (intervention) group and the control group at study endpoint
changes in levels of blood lipids | 3 months
  detection of significant differences in the concentration of fasting total cholesterol (mg/dL), low density lipoprotein (mg/dL), high density lipoprotein (mg/dL), triacyglycerols (mg/dL) between the CDSS (intervention) group and the control group at study endpoint
change in body weight (kg) | 3 months
  significant decrease of body weight (kg) in the CDSS (intervention) group compared to control group at study endpoint
change in body fat mass (%) | 3 moths
  significant decrease of body fat mass (%) in the CDSS (intervention) group compared to control group at study endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Panos Papandreou, Athens, Greece